CLINICAL TRIAL: NCT01617356
Title: Treatment of Temporomandibular Dysfunction With Hypertonic Dextrose Injection: A Randomised Clinical Trial of Efficacy
Brief Title: Treatment of Temporomandibular Dysfunction With Hypertonic Dextrose Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frusso, Ricardo, M.D. (Individual)
Collaborators: Zarate, Miguel, M.D. (Individual)
Responsible Party: Principal Investigator, Ricardo D Frusso, M.D., Principal Investigator, Frusso, Ricardo, M.D.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Buenos Aires 1969
Record Dates: First submitted 2012-06-05; First posted 2012-06-12 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Temporomandibular Joint Disorders
Keywords: TMD; temporomandibular; dextrose; prolotherapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Glucose; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dextrose Injection (Active Comparator)
  Interventions: Other: Injection of 20% dextrose/ 0.2% lidocaine
- Sterile Water Injection (Active Comparator)
  Interventions: Other: Injection of 1 ml of 0.8 SW/0.2% lidocaine

INTERVENTIONS:
Other: Injection of 20% dextrose/ 0.2% lidocaine — Injection at 0, 1, and 2 months of 1 ml of a solution consisting of 20% dextrose and 0.2% lidocaine.
  Arms: Dextrose Injection
Other: Injection of 1 ml of 0.8 SW/0.2% lidocaine — Injection at 0, 1, and 2 months of 1 ml of a solution consisting of 0.8 sterile water and 0.2% lidocaine.
  Arms: Sterile Water Injection

SUMMARY:
Dysfunction of the jaw, associated with pain in the jaw or about the jaw in the face can be quite long lasting and debilitating. Dextrose injection with a small needle has be notably helpful in preliminary studies in reducing pain and improving jaw function. This randomized trial will compare dextrose injection with saline injection for temporomandibular(jaw) dysfunction, also known as TMD.

DETAILED DESCRIPTION:
Longitudinal studies of subjects with temporomandibular dysfunction show a general pattern of symptom diminishment, especially in the elderly. However studies out to 2-8 years show residual symptoms in many and nearly 25% with unabated symptoms. Dextrose injection has been utilized empirically for many years and a marked reduction in pain and luxation after intraarticular and pericapsular dextrose injection has been reported in a recent RCT. However, small study size and lack of a non injection control have prevented any definitive conclusions as the additional efficacy of including dextrose in the injectate. The mechanism of action of dextrose injection was originally thought to be via a brief stimulation of the inflammatory cascade with resultant production of growth factors. However, non-inflammatory dextrose effects on growth factor production have been demonstrated, and, more recently, dextrose has been found to treat neurogenic inflammation (pain from upregulation of the TRPV1 receptor on peptidergic nerves). This has the theoretical benefit of reducing pain, regardless of the status and position of the intraarticular cartilage or degree of degenerative change of the TMD. The primary goal of this study is to evaluate the ability of dextrose injection versus saline injection to reduce pain and improve functional complaints referable to the temporomandibular joint.

ELIGIBILITY:
Inclusion Criteria:

* Facial Pain NRS rating > 5/10
* Jaw symptom rating > 5/10
* Jaw function issues seen on examination

Exclusion Criteria:

* Any potential acute dental issue
* Rheumatic inflammatory disease
* Chronic intake of NSAIDs or corticosteroids.
* Pain in other body location worse than jaw pain
* Pain 10/10 in other body location.

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 3 months in a 0-10 Numerical Rating Scale (NRS) for Jaw Pain | 3 months
  Anchors include "0 = no pain" and "10 = worst pain imaginable" An improvement is a reduction in the NRS scale.
50% or more improvement in 0-10 Numerical Rating Scale (NRS) for Jaw pain from baseline to 3 months | 3 months
  Anchors include "0 = no pain" and "10 = worst pain imaginable." A 50% reduction in the 0-10 NRS is a clinically important outcome.
Change from baseline to 3 months in a 0-10 Numerical Rating Scale (NRS) for jaw dysfunction. | 3 months
  Anchors include "0 = no pain" and "10 = worst pain imaginable" An improvement is a reduction in the NRS scale.
50% or more improvement in 0-10 Numerical Rating Scale (NRS) for for jaw dysfunction to 3 months | 3 months
  Anchors include "0 = no pain" and "10 = worst pain imaginable." A 50% reduction in the 0-10 NRS is a clinically important outcome.
Change from baseline to 1 year in a 0-10 Numerical Rating Scale (NRS) for jaw pain | 1 year
  Anchors include "0 = no pain" and "10 = worst pain imaginable" An improvement is a reduction in the NRS scale.
50% or more improvement in 0-10 Numerical Rating Scale (NRS) for for jaw pain from baseline to 1 year | 1 year
  Anchors include "0 = no pain" and "10 = worst pain imaginable." A 50% reduction in the 0-10 NRS is a clinically important outcome.
Change from baseline to 1 year in a 0-10 Numerical Rating Scale (NRS) for Jaw Dysfunction | 1 year
  Anchors include "0 = no pain" and "10 = worst pain imaginable" An improvement is a reduction in the NRS scale.
50% or more improvement in 0-10 Numerical Rating Scale (NRS) for for jaw dysfunction from baseline to 1 year | 1 year
  Anchors include "0 = no pain" and "10 = worst pain imaginable." A 50% reduction in the 0-10 NRS is a clinically important outcome.

SECONDARY OUTCOMES:
Change in mouth opening in millimeters from baseline to 3 months as manually measured by a Therabite. | 3 months
  An increase in mouth opening in millimeters is considered an improvement in this study.
Satisfaction to 3 months as measured by a 0-10 Numerical Rating Scale (NRS) | 3 months
  Anchors include "0 = no satisfaction" and "10 = complete satisfaction"

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo D Frusso, M.D., Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Zarate MA, Frusso RD, Reeves KD, Cheng AL, Rabago D. Dextrose Prolotherapy Versus Lidocaine Injection for Temporomandibular Dysfunction: A Pragmatic Randomized Controlled Trial. J Altern Complement Med. 2020 Nov;26(11):1064-1073. doi: 10.1089/acm.2020.0207. Epub 2020 Aug 11. PMID 32780636